CLINICAL TRIAL: NCT02751619
Title: Preventive Application Of Lidocaine Patch In Adjunction To Intravenous Morphine Analgesia For Management Of Post-Thoracotomy Pain: Results Of A Randomized, Double Blind, Placebo Controlled Study
Brief Title: Preventive Skin Analgesia With Lidocaine Patch 5% for Controlling Post-thoracotomy Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Campania Luigi Vanvitelli (Other)
Responsible Party: Principal Investigator, Alfonso Fiorelli, MD, PhD, University of Campania Luigi Vanvitelli
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 436/2012
Record Dates: First submitted 2016-04-17; First posted 2016-04-26 (Estimated); Last update posted 2016-04-26 (Estimated); Status verified 2016-04

CONDITIONS: Pain, Postoperative
Keywords: Pre-emptive analgesia; Post-thoracotomy pain; Lidocaine patch
MeSH Terms: conditions — Pain, Postoperative | interventions — Lidoderm

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Lidocaine Group (Experimental): Lidocaine patch 5% (Lidoderm®, Endo Pharmaceuticals Inc, Malvern, PA, USA) measuring 10 x 14 cm and containing 700 mg of Lidocaine, was applied to cover the planned skin incision, marked with a pen by surgeon. Patch was applied for 12 hours during the night, removed for the subsequent 12 hours during the day, and then a new patch was applied at the same level the night after. This process was continued for 3 days before thoracotomy
  Interventions: Drug: Lidocaine patch 5%
- Placebo Patch (Active Comparator): A patch, that was identical in appearance to the active patch but did not contain Lidocaine, was applied to cover the planned skin incision, marked with a pen by surgeon. Patch was applied for 12 hours during the night, removed for the subsequent 12 hours during the day, and then a new patch was applied at the same level the night after. This process was continued for 3 days before thoracotomy
  Interventions: Drug: Placebo patch

INTERVENTIONS:
Drug: Lidocaine patch 5% — Lidocaine patch 5% was applied to cover the planned skin incision for 12 hours during the night and then was removed for the subsequent 12 hours during the day. This process was continued for 3 days before thoracotomy
  Other Names: Lidoderm® (Endo Pharmaceuticals Inc, Malvern, PA, USA)
  Arms: Lidocaine Group
Drug: Placebo patch — A patch without lidocaine was applied to cover the planned skin incision for 12 hours during the night and then was removed for the subsequent 12 hours during the day. This process was continued for 3 days before thoracotomy
  Arms: Placebo Patch

SUMMARY:
Thoracotomy is one of the most painful surgical incision. Uncontrolled acute post-thoracotomy pain reducing deep breathing exercises and secretion clearance increased the incidence of postoperative pulmonary complications including atelectasis, hypoxemia, and postoperative pulmonary infections. Thus, an effective analgesia is crucial in order to reduce perioperative morbidity and hospitalization time and also to prevent chronic post-thoracotomy pain.

Thoracic epidural analgesia and thoracic paravertebral analgesia are currently the standard strategies for thoracic surgery but the difficult of performing them in all patients and their potential complications are all factors that limit their use. Systemic administration of opioids is the simplest and common strategy to provide analgesia but it may be associated with several undesirable effects, such as respiratory depression, sedation, nausea, constipation and vomiting.

In the recent years, preventive analgesia is become one of the most promising strategy of postoperative pain control. It is based on the concept of administering analgesic drugs before the occurrence of nociceptive input in order to prevent central sensitization. The efficacy of preemptive analgesia is unclear and there is no a consensus on its efficacy on controlling pain after thoracic procedure.

Pain following thoracotomy has a multifactorial genesis including surgical incision, intercostal nerve injury, pleural inflammation, and damage of pulmonary parenchyma and of diaphragm. Thus, a multimodal analgesia that intercepts the signalizing at numerous locations could be more effective than a single strategy targeting one site along the pain pathway.

Thus, in the present study, the clinical hypothesis was that the preemptive analgesia of the skin using a new tool as the Lidocaine patch 5% would improve the analgesic effects of systemic morphine analgesia for controlling post-operative pain following thoracotomy.

DETAILED DESCRIPTION:
This was an unicenter, double-blinded, placebo controlled, parallel-group, prospective study conducted at Thoracic Surgery Unit and Anesthesia and Intensive Care Unit of Second University of Naples from January 2013 to May 2015.

All consecutive patients undergoing undergoing anatomical resection by standard lateral thoracotomy for treatment of non small cell lung cancer (NSCLC) were randomly assigned to Lidocaine or Placebo group in 1:1 ratio and no changes to methods after trial commencement as type of randomization or eligibility criteria were attended.

For patients assigned to active group, Lidocaine patch 5% (Lidoderm®, Endo Pharmaceuticals Inc, Malvern, PA, USA) measuring 10 x 14 cm and containing 700 mg of Lidocaine, was applied to cover the planned skin incision, marked with a pen by surgeon. Patch was applied for 12 hours during the night, removed for the subsequent 12 hours during the day, and then a new patch was applied at the same level the night after. This process was continued for 3 days before thoracotomy. In the control group, a placebo patch, that was identical in appearance to the active patch but did not contain Lidocaine, was applied in the same manner for the same time. The pain service, surgical team, and patients were all blinded to treatment group assigned.

All patients received the same anesthetic protocol. All operations were performed in the early morning just after that the patch was removed. The general anesthesia was inducted with i.v. midazolam 0.05 mg/kg, i.v. fentanyl 1-1.4 µg/Kg, i.v. propofol 2.5 mg/kg, i.v. and rocuronium bromide 0.6 mg/kg. The patient was maintained with desflurane 4-6%, sulfentanil 0.5-1 micro/Kg, rocuronium bromide 0.6-0.8 mg/Kg, based on heart rate and blood pressure stability. A selective ventilation was performed with a double-lumen endobronchial tube in all cases and no additional analgesics were injected during surgery.

All patients had the same length of skin incision and a standard muscle-sparing lateral thoracotomy. The latissimus dorsi muscle and the underlying serratus anterior muscle were spared and the chest was entered over the top of the unresected and unshingled sixth rib. A standard Finocchietto chest retractor was then placed and slowly opened to avoid rib fracture. After completion of the appropriate anatomical lung resection, a single 28 F chest drainage was systematically placed in pleural cavity. The same chest closure was performed in all patients in a standard manner using intracostal sutures.

Patient was extubated in the operating room and transferred to the surgical ward. The postoperative analgesia was performed with intravenous morphine administered through Patient Controlled-Analgesia (Automed 3300, AceMedical Co.) delivery. Morphine 1 mg was given for each request and continuous infusion was at a rate of 1 mg/h. Both groups had a 10 min lockout period and a safe higher limit of 20 mg in 4 hours. If VAS scores exceeded 4/10 scores, rescue analgesia was intravenously administered according to a standardized institutional protocol for pain treatment until the pain was relieved to a level falling below a VAS score < 4. Patient Controlled Analgesia (PCA) was continued for up to 2 days, until patients could tolerate oral opioid medications and/or anti-inflammatory analgesics. However, these medications were not considered in the analysis.

The intergroup differences were assessed in order to evaluate whether the pre-emptive analgesia obtained with Lidocaine patch would have effects on pain scores (primary end-point), consumption of analgesics, recovery of respiratory function and peripheral painful pathways (secondary end-points).

ELIGIBILITY:
Inclusion Criteria:

* More than 18 years old
* Anatomical resection by standard lateral thoracotomy for treatment of non small cell lung cancer

Exclusion Criteria:

* Allergy to Lidocaine
* American Society of Anaesthesiologist (ASA) classification score more than 3
* History of previous thoracic surgical procedures and/or of chronic pain or taking regular analgesics
* Pneumonectomy or concomitant decortication and/or chest wall injury or resection,
* Psychiatric illness
* Participation to other studies

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2013-01; Primary Completion 2015-05 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Changes in Pain Score measured with Visual Analogue Scale at rest and after coughing | Post-operative follow-up-points: 6 hours, 12 hours , 24 hours , 36 hours, 48 hours and 72 hours
  10-score Visual Analogue Scale (VAS) ranging from 0=absence of pain to 10= maximal level of pain

SECONDARY OUTCOMES:
The frequency for hour of activation of PCA Device | Post-operative follow-up: 6 hours; 6-12 hours; 12- 24 hours; 24-36 hours, and 36-48 hours.
  The sum of the frequency of activation of PCA system
Morphine consumption | Post-operative follow-up: 6 hours; 6-12 hours; 12- 24 hours; 24-36 hours, and 36-48 hours.
  The total morphine consumption expressed (the sum of additional intravenous morphine bolus infusions and the morphine delivered by the PCA system)
Flow Expiratory Volume in one second (FEV1%) | Post-operative follow-up: 72 hours; 96 hours; 120 hours
  The best of three efforts measured with a spirometer was used for the analysis.
Forced Vital Capacity (FVC%) | Post-operative follow-up: 72 hours; 96 hours; 120 hours
  The best of three efforts measured with a spirometer was used for the analysis.
Laser Evoked Potential Tests. | Follow-up: 1 month, 3 months, and 6 months after operation
  Laser stimulation, delivered by Nd:YAG (neodymium-doped yttrium aluminium garnet (Nd:YAG) laser, was applied at level of thoracotomy scar, the main territory corresponding to the distribution of pain. The results were evaluated for amplitude and latency differences between the vertex negativity (N2) appearing around 240 ms and the following positivity (P2) appearing around 360 ms after stimulus onset.

CONTACTS AND LOCATIONS:
Overall Officials: Mario Santini, MD, Study Chair — University of Campania Luigi Vanvitelli

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Background] Cerfolio RJ, Bryant AS, Bass CS, Bartolucci AA. A prospective, double-blinded, randomized trial evaluating the use of preemptive analgesia of the skin before thoracotomy. Ann Thorac Surg. 2003 Oct;76(4):1055-8. doi: 10.1016/s0003-4975(03)01023-3. PMID 14529984
- [Background] Garzon-Rodriguez C, Casals Merchan M, Calsina-Berna A, Lopez-Romboli E, Porta-Sales J. Lidocaine 5 % patches as an effective short-term co-analgesic in cancer pain. Preliminary results. Support Care Cancer. 2013 Nov;21(11):3153-8. doi: 10.1007/s00520-013-1948-7. Epub 2013 Sep 3. PMID 24000041
- [Background] Vrooman B, Kapural L, Sarwar S, Mascha EJ, Mihaljevic T, Gillinov M, Qavi S, Sessler DI. Lidocaine 5% Patch for Treatment of Acute Pain After Robotic Cardiac Surgery and Prevention of Persistent Incisional Pain: A Randomized, Placebo-Controlled, Double-Blind Trial. Pain Med. 2015 Aug;16(8):1610-21. doi: 10.1111/pme.12721. Epub 2015 Jul 14. PMID 26176878
- [Background] Habib AS, Polascik TJ, Weizer AZ, White WD, Moul JW, ElGasim MA, Gan TJ. Lidocaine patch for postoperative analgesia after radical retropubic prostatectomy. Anesth Analg. 2009 Jun;108(6):1950-3. doi: 10.1213/ane.0b013e3181a21185. PMID 19448228
- [Background] Cheng YJ. Lidocaine Skin Patch (Lidopat(R) 5%) Is Effective in the Treatment of Traumatic Rib Fractures: A Prospective Double-Blinded and Vehicle-Controlled Study. Med Princ Pract. 2016;25(1):36-9. doi: 10.1159/000441002. Epub 2015 Nov 6. PMID 26539836